CLINICAL TRIAL: NCT03707639
Title: Phase II Study of the Combination of Apatinib and POF (Paclitaxel Plus Oxaliplatin Plus 5-fluorouracil Plus Leucovorin)
Brief Title: Study of the Combination of Apatinib and POF
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FNF011
Record Dates: First submitted 2018-10-12; First posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Gastric Adenocarcinoma
MeSH Terms: interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Apatinib plus POF (Experimental): Apatinib (500 mg qd p.o.) plus POF until disease progression or intolerable toxicity or refused by the patients.
  Interventions: Drug: Apatinib; Drug: POF

INTERVENTIONS:
Drug: Apatinib — Apatinib (500 mg qd p.o.) until disease progression or intolerable toxicity or refused by the patients.
Drug: POF — The POF regimen consisted of a 3-hour infusion of paclitaxel (135 mg/m2) followed by oxaliplatin (85 mg/m2) and Calcium Levofolinate (200 mg/m2).Subsequently, a 46-hour infusion of fluorouracil (2400 mg/m2) was administered using an ambulatory pump, repeating the cycle every 14 days.

SUMMARY:
In previous studies, we found that POF (A combination of oxaliplatin, fluorouracil and Paclitaxel) regimen appears to be of good efficacy and is well tolerated in patients with advanced gastric cancer. Apatinib is an orally antiangiogenic agent. It was approved and launched in China in 2014 as a 3rd-line treatment for patients with advanced gastric cancer. Therefore, investigators conducted the dose escalation phase I study to explore the safety of combination of apatinib and POF as first-line treatment for advanced gastric cancer. Now we are going to start a phase 2 trial with apatinib 500mg + POF as first-line therapy to investigate the efficacy and safety in the patients with advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

Patients with advanced unresectable, histologically confirmed adenocarcinoma of the gastric or gastroesophageal junction.

No previous treatment with chemotherapy or radiation therapy. Ability to take medications orally. With measurable lesions. Patients must have a performance status of 0-1 on the Eastern Cooperative Oncology Group (ECOG) scale.

Without serious system dysfunction and could tolerate chemotherapy. With normal marrow, liver and renal function: a hemoglobin (HGB) of ≥100g/L (without blood transfusion during 14 days); a leucopenia count of ≥4.0×109/L; a platelet count of ≥100×109/L; a total bilirubin (TBil) of ≤1.5 upper normal limitation (UNL); a creatinine (Cr) of ≤ 1.5 UNL; a creatinine clearance rate ≥ 50ml/min (Cockcroft-Gault); a alanine aminotransferase (ALAT) and aspartate aminotransferase (ASAT) of ≤2.5 UNL or ≤5 UNL in case of liver metastasis.

Life expectancy ≥3 months. With normal electrocardiogram results and no history of congestive heart failure.

Without bleeding and thrombosis disease. With normal coagulation function: activated partial thromboplastin time (APTT), prothrombin time (PT) and INR, each ≤ 1.5 x ULN.

Female subjects of child-bearing potential must agree to use contraceptive measures starting 1 week before the administration of the first dose of apatinib until 8 weeks after discontinuing study drug. Male subjects must agree to use contraceptive measures during the study and 8 weeks after last dose of study drug With written informed consent signed voluntarily by patients themselves or their supervisors witted by doctors.

With good compliance and agree to accept follow-up of disease progression and adverse events.

Exclusion Criteria:

Patients with a history of another neoplastic disease within the past three years, excluding basal cell carcinoma of the skin, cervical carcinoma in situ, or nonmetastatic prostate cancer.

Patients with brain or central nervous system metastases, including leptomeningeal disease.

Pregnant (positive pregnancy test) or breast feeding. Serious, non-healing wound, ulcer, or bone fracture. Significant cardiac disease as defined as: unstable angina, New York Heart Association (NYHA) grade II or greater, congestive heart failure, history of myocardial infarction within 6 months Evidence of bleeding diathesis or coagulopathy.

History of a stroke or CVA within 6 months. Clinically significant peripheral vascular disease. Inability to comply with study and/or follow-up procedures. Patients with any other medical condition or reason, in that investigator's opinion, makes the patient unstable to participate in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | From enrollment to 3 months after treatment
  According to RECIST 1.1

SECONDARY OUTCOMES:
Progression-free survival | From enrollment to progression of disease. Estimated about 12 months.
  The length of time from enrollment until the time of progression of disease
Overall survival | From enrollment to death of patients. Estimated about 18 months
  The length of time from enrollment until the time of death
Toxicity According to NCI CTCAE 4.03 criteria | From enrollment to 3 months after treatment
  According to NCI CTCAE 4.03 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Rongbo Lin, Study Chair — Fujian Cancer Hospital
Locations (1):
- Rongbo Lin, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No